CLINICAL TRIAL: NCT03725358
Title: A Cluster-randomized Controlled Trial to Increase the Uptake of Long-acting Reversible Contraceptives Among Adolescent Females and Young Women in Cameroon
Brief Title: A Cluster-RCT to Increase the Uptake of LARCs Among Adolescent Females and Young Women in Cameroon.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Problems with the Performance-Based Financing System in Cameroon, combined with the restrictions on movement brought on by the Covid-19 pandemic.
Sponsor: World Bank (Other)
Collaborators: Stanford University (Other); George Washington University (Other); University of Exeter (Other); University of California, San Diego (Other); Yaounde Gynecology, Obstetrics and Pediatrics Hospital (Unknown)
Responsible Party: Principal Investigator, Berk Ozler, Principal Investigator, World Bank
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: LARCs-2019
Record Dates: First submitted 2018-10-29; First posted 2018-10-31 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Contraception Behavior; Contraceptive Usage; Contraceptive Method Switching; Contraception
Keywords: adolescent sexual and reproductive health, maternal mortality, teen pregnancy, LARCs
MeSH Terms: conditions — Contraception Behavior; Maternal Death | interventions — Amyloid

STUDY DESIGN:
Intervention Model Description: three supply-side interventions (including control condition) are being crossed with three levels of subsidies for LARCs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Control: no training, low subsidies (Experimental): No provider training and low (status quo) subsidies received: business as usual
  Interventions: Behavioral: Control
- No training, medium-level subsidies (Experimental): No provider training, but receiving medium-level PBF payments for contraceptive methods provided
  Interventions: Behavioral: Control
- No training, high-level subsidies (Experimental): No provider training, but receiving high-level PBF payments for contraceptive methods provided
  Interventions: Behavioral: Control
- Training, low-level subsidies (Experimental): Providers being trained on modern contraception, but receiving low-level (status quo) PBF payments for contraceptive methods provided
  Interventions: Behavioral: Training
- Training, medium-level subsidies (Experimental): Providers being trained on modern contraception, but receiving medium-level (status quo) PBF payments for contraceptive methods provided
  Interventions: Behavioral: Training
- Training, high-level subsidies (Experimental): Providers being trained on modern contraception, but receiving high-level (status quo) PBF payments for contraceptive methods provided
  Interventions: Behavioral: Training
- Training+App, low-level subsidies (Experimental): Providers being trained on modern contraception and receiving a tablet-based decision-support tool (app), but receiving low-level (status quo) PBF payments for contraceptive methods provided
  Interventions: Behavioral: App
- Training+App, medium-level subsidies (Experimental): Providers being trained on modern contraception and receiving a tablet-based decision-support tool (app), but receiving medium-level (status quo) PBF payments for contraceptive methods provided
  Interventions: Behavioral: App
- Training+App, high-level subsidies (Experimental): Providers being trained on modern contraception and receiving a tablet-based decision-support tool (app), but receiving high-level (status quo) PBF payments for contraceptive methods provided
  Interventions: Behavioral: App

INTERVENTIONS:
Behavioral: Training — Health facilities assigned to this group will receive a two-week training intervention on modern contraceptive methods and counseling techniques - aimed at nurses conducting family planning services. This new curriculum was developed by a large group of experts convened by the Ministry of Health in February 2018. The cascade training that is developed by the national government (cascading down to regions, districts, and finally health facilities) is a 15-day training module that targets family planning nurses, covering theory, practical knowledge (practicing administrations and removals), and counseling of clients.
  Arms: Training, high-level subsidies; Training, low-level subsidies; Training, medium-level subsidies
Behavioral: App — Health facilities assigned to this group will receive the same programming as the facilities in S1, but they will also be provided with tablets equipped with the "job aid," which subsumes the basic data collection software used by the remaining facilities. They will also receive additional training on the use of the tablet-based "job aid."
  The "app" is a tablet-based decision-support tool, which is designed for use by the family planning nurse conducting counseling sessions and records the answers to a series of questions that elicit the client's life goals, fertility plans, needs, and preferences regarding contraceptive methods, as well as her medical eligibility (birth history, pregnancy check, breastfeeding status, blood pressure, medications, etc.).
  Arms: Training+App, high-level subsidies; Training+App, low-level subsidies; Training+App, medium-level subsidies
Behavioral: Control — The comparison group includes facilities that continue business as usual (no FP training or tablet-based job aid). Each facility in this group will receive a tablet equipped with basic data collection software and a one-day training to use the tablets.
  Arms: Control: no training, low subsidies; No training, high-level subsidies; No training, medium-level subsidies

SUMMARY:
The study investigators propose to test various supply-side approaches to increase the numbers of both SARCs (short-acting reversible contraceptives, i.e. the pill and injectable) and especially LARCs (long-acting reversible contraceptives, i.e. the IUD and implant) administered by health facilities to reproductive-age females in Cameroon, particularly adolescents who may be unmarried and/or nulliparous. The study investigators will do this via interventions at primary health facilities, which include training of providers on family planning; the introduction of a tablet-based decision support tool for counseling women on family planning; and increased subsidies for LARCs within the performance-based financing (PBF) system. This approach is expected to benefit the population directly by decreasing maternal mortality and undesired pregnancies and indirectly by reducing side effects that arise due to current one-size-fits-all FP (family planning) counseling; improving the health of children due to improved birth spacing; and increasing human capital accumulation among children and young (often school-age) potential mothers.

ELIGIBILITY:
Inclusion Criteria:

* Facilities in the East Region of Cameroon providing family planning services under the performance-based financing (PBF) system.

Exclusion Criteria:

* Facilities that have not administered any modern contraceptive methods in the past quarter

Ages: 10 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
The total number of modern contraceptives (SARCs + LARCs) administered per facility per quarter | 12 months
The total number of LARCs administered per facility per quarter | 12 months

SECONDARY OUTCOMES:
The total number of counseling sessions conducted per facility per quarter | 12 months
Prices charged for LARCs and SARCs per quarter | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Berk Ozler, PhD, Principal Investigator — World Bank

IPD SHARING:
Plan to Share IPD: Undecided
We will likely share de-identified anonymous participant data publicly after the trial ends and our analyses are completed.